CLINICAL TRIAL: NCT07165262
Title: Effect of Different Anesthetic Drugs on Electrocorticography (ECOG), Randomized Controlled Double-blinded Study
Brief Title: Effect of Different Anesthetic Drugs on Electrocorticography (ECOG).
Acronym: ECOG-Anaes
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Cancer Hospital Egypt 57357 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: N-0061-008-025
Record Dates: First submitted 2025-08-24; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Epilepsy; Brain Tumor
Keywords: ECOG, Brain Tumors, Ketamine, Fentanyl
MeSH Terms: conditions — Epilepsy; Brain Neoplasms | interventions — Fentanyl; Ketamine

STUDY DESIGN:
Intervention Model Description: Signed consent will be obtained from all patient's guardian after a detailed preoperative explanation. 88 pediatric patients aged 2-18 years with brain tumor for excision with aid of ECOG and American Society of Anesthesiologist physical status II-III.
  Patients will be divided into two groups computer-allocated, given fentanyl (1ug/kg) and Ketamine (0.5mg/kg) for spike stimulation.
  Patients, anesthesiologists, surgeons, and neurophysiologist will be blinded to the group allocation of patients throughout the study.
  Spike frequency and waveform (pre-, during, and post-excision) intraoperatively will be recorded by the neurophysiologist which will be proportionate directly to the state of stimulation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fentanyl (Active Comparator): fentanyl will be used as bolus (1 µg/kg) for spike stimulation
  Interventions: Drug: Fentanyl (IV)
- Ketamine (Experimental): ketamine will be used (0.5 mg/kg) for spike stimulation
  Interventions: Drug: Ketamine (0.5 mg/kg)

INTERVENTIONS:
Drug: Fentanyl (IV) — Fentanyl, Intravenous bolus administration at a dose of 1 microgram per kilogram of body weight administered once before spike stimulation and another time after resection of epileptic foci for spike stimulation.
  Other Names: fentanyl citrate
  Arms: Fentanyl
Drug: Ketamine (0.5 mg/kg) — Ketamine, Intravenous bolus administration at a dose of 0.5 milligram per kilogram of body weight administered once before spike stimulation and another time after resection of epileptic foci for spike stimulation.
  Other Names: ketamine hydrochloride
  Arms: Ketamine

SUMMARY:
Prospective, double-blind, randomized-controlled study for pediatric cases scheduled for brain tumor excision with the aid of electrocorticography (ECOG). Intraoperative ECOG has been used in an effort to localize the site of epileptogenicity through the demonstration of Interictal Epileptiform Discharges (IED) persistence, frequency, and distribution. During ECOG, pharmaco-activation may be required in order to activate Interictal Epileptiform Abnormalities (IEAs). Frequency of IEAs will be measured for each drug.

The effects of anesthetic agents on intraoperative ECOG, as we assume that fentanyl will be superior to ketamine.

DETAILED DESCRIPTION:
Brain tumors can be responsible for epilepsy refractory to medical therapy. These are typically slow-growing tumors, and surgery aims to cure the patient's seizure disorder. One of the main uses of electrocorticography is mapping the cortical regions associated with epileptiform activity. This information is used to plan resection boundaries. Electroencephalography (EEG) electrodes are placed directly on the cortical surface, and epileptiform activity is identified, and this can guide the extent of resection. This technique is referred to as intraoperative electrocorticography (IOECOG).

IOECOG has been used to localize the site of epileptogenicity through the demonstration of Interictal Epileptiform Discharges (IED) persistence, frequency, and distribution. As the intraoperative time is short, clinical seizures are usually not captured by ECOG, but the presence and location of IEAs can be used to localize the epileptogenic focus and guide the resection.

During ECOG, pharma coactivation may be required to activate IEAs. Fentanyl and ketamine can be used for this

ELIGIBILITY:
Inclusion Criteria:

* Age (2-18) Years scheduled for brain tumor excision with aid of ECOG
* ASA physical status (II-III).
* Patient undergoing brain surgery with epileptic focus.

Exclusion Criteria:

* guardian refusal.
* Patients with hypertension, ischemic heart disease, arrhythmia, or respiratory or renal dysfunction.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 88 (Actual)
Dates: Start 2025-08-18 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Effect of fentanyl and ketamine on frequency of spike activation during intraoperative ECOG | 18 months
  The frequency of spikes will be recorded at baseline (before using the drug) and after using the drug before resection. After resection of the epileptic foci, restimulation with the drug will be done and spikes will be recorded.
Effect of fentanyl and ketamine on amplitude of the spikes activated during intraoperative ECOG. | 18-month
  The amplitude of spikes will be recorded at baseline (before using the drug) and after using the drug before resection. After resection of the epileptic foci, restimulation with the drug will be done, and the spike amplitude will be recorded.
Effect of fentanyl and ketamine on number of leads with activated spikes during intraoperative ECOG. | 18-months
  The number of leads with activated spikes will be recorded at baseline (before using the drug) and after using the drug before resection. After resection of the epileptic foci, restimulation with the drug will be done, and the number of leads with activated spikes will be recorded.

SECONDARY OUTCOMES:
The effect of fentanyl and ketamine on blood pressure is to be measured with the drug administered for stimulation. | 18 months
  The effect of fentanyl and ketamine on blood pressure will measured pre- and post-drug administration.
The effect of fentanyl and ketamine on heart rate is to be measured with the drug administered for stimulation. | 18-month
  The effect of fentanyl and ketamine on heart rate will be measured pre- and post-drug administration.
The effect of fentanyl and ketamine on recovery time. | 18 month
  The effect of fentanyl and ketamine on recovery time will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Suzan A. Abdelrahman, consultant, Principal Investigator — Children's Cancer Hospital Egypt 57357
Locations (2):
- Egypt (2):
  - Children's Cancer Hospital Egypt 57357, Cairo
  - Children Cancer Hospital 57357, Cairo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lemieux, L., et al. (2012). "Invasive EEG for Epilepsy Surgery: Current Techniques and Considerations." Journal of Clinical Neurophysiology, 29(3), 246-257.